CLINICAL TRIAL: NCT00483002
Title: Post Marketing Surveillance Study To Observe Safety And Efficacy Of Champix® Tablets
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3051083
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Results first posted 2012-05-11 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-04

CONDITIONS: Smoking Cessation
Keywords: A prospective and observational program to monitor use in real practice including efficacy of Varenicline in Korea.
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy smokers
  Interventions: Drug: varenicline

INTERVENTIONS:
Drug: varenicline — As prescribed by physician in usual clinical practice.
  Other Names: Champix, Chantix, CP-526,555

SUMMARY:
To monitor use in real practice including safety and efficacy of Champix tablets 0.5mg, 1mg medication for 12 weeks in smokers

DETAILED DESCRIPTION:
No sampling method will be applied to this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects selected for this study are those who would have been prescribed Champix tablets by the physician according to the subject's condition in usual clinical practice.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy smokers
Sampling Method: Non-Probability Sample
Enrollment: 3719 (Actual)
Dates: Start 2007-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Ock M, Shin JS, Ra SW. Safety and Effectiveness of Varenicline in Korean Smokers: A Nationwide Post-Marketing Surveillance Study. Patient Prefer Adherence. 2022 Feb 15;16:413-426. doi: 10.2147/PPA.S344757. eCollection 2022. PMID 35210758
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051083&StudyName=Post%20Marketing%20Surveillance%20Study%20To%20Observe%20Safety%20And%20Efficacy%20Of%20Champix%AE%20Tablets

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: Varenicline tartrate tablets 0.5 milligram (mg) or 1 mg administered as per investigator's discretion for 12 weeks.
Period: Overall Study
Arm/Group | Varenicline
Started | 3719
Completed | 1165
Not Completed | 2554
Not completed — Adverse Event | 68
Not completed — Lack of Efficacy | 555
Not completed — Lost to Follow-up | 962
Not completed — Other | 2
Not completed — Other | 967

BASELINE CHARACTERISTICS:
Arm/Group | Varenicline
Number analyzed (Participants) | 3719
Age Continuous [Mean (Standard Deviation); unit: Years] | 49.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 340
  Male | 3379

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 7-day Point Prevalence From Week 3 to Less Than Week 7
Description: Treatment effectiveness was measured by 7-day point prevalence of smoking abstinence status. The smoking status was categorized as smoking or abstained smoking based on 2 parameters: if participant smoked any cigarettes (even a puff) in the last 7 days (Yes/No); if participant used any other nicotine-containing products in the last 7 days (Yes/No).
Time Frame: Week 3 through Week 7
Population: Study population included all those participants who received the study medication more than once and were available for follow up. Here, the 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Varenicline
Number analyzed (Participants) | 2922
Percentage of participants | 59.55 [57.77 to 61.33]

2. Primary Outcome: Percentage of Participants With 7-day Point Prevalence From Week 7 to Less Than Week 11
Description: as for outcome 1
Time Frame: Week 7 through Week 11
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Varenicline
Number analyzed (Participants) | 1520
Percentage of participants | 73.29 [71.07 to 75.51]

3. Primary Outcome: Percentage of Participants With 7-day Point Prevalence for at Least Week 11
Description: as for outcome 1
Time Frame: At least Week 11
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Varenicline
Number analyzed (Participants) | 1449
Percentage of participants | 77.02 [74.85 to 79.18]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Varenicline
Serious Adverse Events (participants affected / at risk) | 4/3719
Other Adverse Events (participants affected / at risk) | 342/3719
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=3719)
Pneumonia (Infections and infestations) | 1
Cerebral artery stenosis (Nervous system disorders) | 1
Neuritis (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Thinking abnormal (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=3719)
Appetite decreased/anorexia (General disorders) | 7
Fatigue/malaise/adynamia (General disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 13
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 12
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 30
Epigastric discomfort (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival oedema (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 191
Vomiting (Gastrointestinal disorders) | 9
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Increased appetite (Metabolism and nutrition disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 5
Dreamy state (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 26
Mental impairment (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 9
Abnormal dreams (Psychiatric disorders) | 30
Depression (Psychiatric disorders) | 8
Hallucination (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 29
Nightmare (Psychiatric disorders) | 6
Sleep disorder (Psychiatric disorders) | 14
Suicidal ideation (Psychiatric disorders) | 1
Nipple pain (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Planned observation time points at 4, 8 and 12 weeks were reported as from week 3 to less than week 7, from week 7 to less than week 11, at least week 11. As this is non-interventional study it is likely that adverse events had been under reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.